CLINICAL TRIAL: NCT04926974
Title: Community Access Through Remote Eyesight (CARE) Study
Acronym: CARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New England College of Optometry (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency); University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CARE
Record Dates: First submitted 2021-06-02; First posted 2021-06-15 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Low Vision
MeSH Terms: conditions — Vision, Low

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Seeing AI Smart Phone App (Experimental): Intervention: Behavioral: Low Vision Rehabilitation
  Interventions: Behavioral: Low Vision Rehabilitation
- Supervision+ Smart Phone App (Experimental): Intervention: Behavioral: Low Vision Rehabilitation
  Interventions: Behavioral: Low Vision Rehabilitation
- Aira Smart Phone App (Experimental): Intervention: Behavioral: Low Vision Rehabilitation
  Interventions: Behavioral: Low Vision Rehabilitation

INTERVENTIONS:
Behavioral: Low Vision Rehabilitation — Smart phone App

SUMMARY:
Study is a randomized clinical trial evaluating the efficacy of novel mobile application technologies (including Seeing AI, Aira, and Supervision+) to improve quality of life in older adults with low vision by expanding community access and providing assistance with activities of daily living. Aira provides real-time remote personal assistance through a sighted Aira agent supplying direct feedback to assist with visual tasks. Seeing AI provides optical character recognition allowing any text to be read aloud, color identification, bar code reading, scene description, and facial recognition based on stored photos. Supervision + allows one to use the phone as a magnifier, providing magnification and contrast enhancement using the camera of the mobile phone. This study seeks to understand the potential of these technologies to improve daily activities, community participation, independence, and self-sufficiency in this group by examining a technological approach, which has not yet undergone rigorous investigation in a diverse population of older adults with visual impairment. Project objectives are to evaluate mobile applications in a wide range of visual disability, categorized into three groups: (1) mild to moderate visual acuity loss, (2) severe to profound visual acuity loss, and (3) legal blindness secondary to visual field loss. Participants are randomized to one of three intervention groups: (1) Supervision+ application, (2) Aira application, or (3) Seeing AI application for a period of 6 months. For the Aira intervention group, participants will be assigned either with 'restricted' access (current open access areas plus 30 minutes/month anywhere), or 'unrestricted' access (700 minutes), for a period of 3 months with a 3 month cross-over period. Participants may elect to continue the study for an additional 3 months during which time they have access to all 3 study mobile applications. Outcome measures include assessment of changes at three, six and nine months post-intervention for: visual ability, health state (including depression), self-efficacy, loneliness, life space, distances travelled from the home, and types of services obtained.

ELIGIBILITY:
Inclusion Criteria:

* age 55 years + (no upper limit)
* reside in CA state (for subjects enrolled at UCLA)
* reside in New England states of MA, NH, CT or RI (for subjects enrolled at NECO)
* best-corrected visual acuity 20/40 to 20/800 in the better eye or visual field diameter less than 20 degrees in the better eye
* English speaking
* Ability to demonstrate proficiency with the smartphone and mobile app at 4 weeks post initial training
* no previous use of the Aira app, Seeing AI app or Super Vision+ app on a smartphone (<5 uses in lifetime)

Exclusion Criteria:

* out of the country for >2 weeks during study intervention period if cannot use their own international data plan on their own phone
* unable to successfully complete the initial on-boarding call for Aira service with an agent as documented by the Aira agent's log (if randomized to Aira)
* schedules not permitting participation in planned study duration (including planning to move or take extended vacation during study period)
* inability to understand study procedures or communicate responses in a consistent manner (cognitive impairment as per TICS)
* substance abuse
* significant hearing loss (unable to hear communication by phone)
* significant medical condition likely to limit participation or lifespan
* participating in another clinical trial that involves treatment that could impact visual function during the study period
* participant in another clinical trial that involves a treatment or intervention that could impact visual functioning
* begins use of a new vision-related app during the trial period for the study

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
Visual ability change score | AI questionnaire will be administered three times over 6 months: baseline, 3-months post-intervention and 6-months post-intervention, and also 9 months post-intervention
  The primary outcome measure is the person change score (before and after intervention), from the adaptive Massof Activity Inventory (AI) Questionnaire. The AI has an item bank of 510 items organized into 50 goals and 460 related visually-based tasks. Subscales range from 0 (not important) to 3 (very important). For those goals rated as important, subjects are asked to rate the task difficulty on subscales of 0 (impossible to do without help) to 5 (not difficult). Rasch analysis is employed to estimate visual ability from these difficulty ratings, on an interval scale. With Rasch analysis person measures are estimated, whereby a more positive person measure reflects greater visual ability.
  In this study, we will explore the the difference in person measures (i.e. change score) after the intervention at 3 and 6 months. A larger, more positive change score indicates greater visual ability since intervention.

SECONDARY OUTCOMES:
Health-related Quality of Life: SF-36 | will be administered three times over 6 months: baseline, 3-months post-intervention and 6-months post-intervention and also 9 months post-intervention
  questionnaire; scale ranges from 1 (excellent) to 5 (poor), with higher values indicating greater difficulty.
Beck Depression Inventory | will be administered three times over 6 months: baseline, 3-months post-intervention and 6-months post-intervention and also 9 months post-intervention
  questionnaire; subscales range from 0 to 3, with higher values indicating greater depression.
Community Living: Life Space Questionnaire | will be administered three times over 6 months: baseline, 3-months post-intervention and 6-months post-intervention and also 9 months post-intervention
  questionnaire; subscales range from 1 (Yes) to 2 (No), with a higher total value indicating a more restricted life space.
3-item UCLA Loneliness Scale | will be administered three times over 6 months: baseline, 3-months post-intervention and 6-months post-intervention and also 9 months post-intervention
  questionnaire; subscales range from 1 to 3, with a high value indicating increased loneliness.
New General Self Efficacy Scale | will be administered three times over 6 months: baseline, 3-months post-intervention and 6-months post-intervention and also 9 months post-intervention
  questionnaire; subscales range from 1 to 5, with a higher value indicating greater self-efficacy.
App usage frequency | at 3 months post-intervention and 6 months post intervention and also 9 months post-intervention
  App usage in minutes.

OTHER OUTCOMES:
Telephone Interview of Cognitive Status (TICS) | administered at time of enrollment
  questionnaire; with subscales 0 to 1, with higher scores indicating greater cognitive ability.
Psychosocial Impact of Assistive Devices Scale (PIADS) | administered at 3-months post-intervention and 6-months post-intervention and also 9 months post-intervention
  questionnaire; with subscales from -3 to 3, higher scores indicate greater affinity of a particular factor to assistive technology use.
Aira Explorer Survey post intervention feedback | 6 months and also 9 months post-intervention
  (specific to those participants randomized to Aira); questionnaire, with subscales ranging from 0 to 10, higher scores indicate stronger agreement or helpfulness of the Aira App.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UCLA Stein Eye Institute, Los Angeles, California
  - New England College of Optometry, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared according to the protocols stipulated by NIDILRR and the IRB at NECO and UCLA.

REFERENCES:
- [Derived] Gobeille M, Bittner AK, Malkin AG, Ho J, Idman-Rait C, Estabrook M, Ross NC; CARE Study Team. Rasch analysis of the new general self efficacy scale: an evaluation of its psychometric properties in older adults with low vision. Health Qual Life Outcomes. 2024 Oct 23;22(1):90. doi: 10.1186/s12955-024-02306-2. PMID 39443965
- [Derived] Bittner AK, Gobeille M, Malkin AG, Ho J, Idman-Rait C, Estabrook M, Ross NC; CARE Study Team. Life space limitations in visually impaired older adults. Optom Vis Sci. 2024 Jun 1;101(6):321-328. doi: 10.1097/OPX.0000000000002150. PMID 38990234
- [Derived] Malkin AG, Bittner AK, Ho J, Idman-Rait C, Estabrook M, Ross NC; CARE Study Team. Factors related to training time and achieving proficiency with visual-assistive mobile applications in visually impaired older adults. Optom Vis Sci. 2024 Jun 1;101(6):351-357. doi: 10.1097/OPX.0000000000002135. Epub 2024 May 31. PMID 38820379